CLINICAL TRIAL: NCT02206451
Title: Assessing Human-to-Mosquito Transmission in Volunteers Participating in Malaria Vaccine Candidate Trials in Don(SqrRoot)(Copyright)gu(SqrRoot)(Copyright)Bougou Mali
Brief Title: Assessing Human-to-Mosquito Transmission in Volunteers Participating in Malaria Vaccine Candidate Trials in Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914159; 14-I-N159
Record Dates: First submitted 2014-07-31; First posted 2014-08-01 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2016-06-29

CONDITIONS: Malaria
Keywords: Assay; Infection; Direct Skin Feed; Midgut; Parasite
MeSH Terms: conditions — Malaria; Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Background:

- Malaria is a disease that affects many people in Mali and in Africa. It is caused by germs that are spread by mosquito bites. Researchers are creating vaccines that they hope will prevent malaria infection and/or the spread of it.

Objective:

- To test if the PfSPZ vaccine can stop malaria spread by mosquitoes.

Eligibility:

- People currently enrolled in the ongoing PfSPZ malaria vaccine trial. Participants must be willing to have uninfected mosquitoes bite them.

Design:

* Participants will be able to take part in this study at every visit after receiving all scheduled vaccinations.
* Participants will be asked whether they are willing to participate in the procedures. Female participants will have a pregnancy test.
* Researchers will put about 60 mosquitoes in 2 or 3 cups (20 or 30 in each cup). They will hold each cup to the participant s leg or arm so the mosquitoes can bite. These mosquitoes do not carry germs and will take about 3 drops of blood total.
* Participants will get a cream for any swelling or itching.
* Participants will be checked the next day for any discomfort.
* Participants may take part in this feeding test multiple times, if they are willing.
* If participants have malaria parasites in their blood, they may be asked to take part in another study. For this, they will sleep alone in their hut the night after the feeding test. A study team will set up nets to collect mosquitoes that may have bitten the participant overnight.

DETAILED DESCRIPTION:
A vaccine which interrupts malaria transmission (VIMT) is a critical tool to achieve the ultimate goal of eradication of this disease. VIMTs work by inducing humoral responses in vaccinated individuals that inhibit the development of malaria parasites in the mosquito, and combined humoral and cellular responses that inhibit the establishment of infection in humans. Overall efficacy of these vaccines is evaluated by measuring reduction of infection and clinical cases among vaccinees and the parasite infectivity to mosquitoes, (human-to-mosquito transmissibility), before and after vaccination, and with or without vaccination. One of the candidate VIMTs, the PfSPZ Vaccine, is currently being tested in Mali for safety, tolerance, and immunogenicity.

The objective of this Feeding Assay Protocol is to explore the effect of the PfSPZ Vaccine, on interrupting human-to-mosquito transmission. Individuals from the the PfSPZ Vaccine trial in 2014 who also consent to be enrolled in this Feeding Assay Protocol will be eligible to participate in procedures including direct skin feeds (DSF) and experimental huts (EH). The human-to-mosquito transmission will be evaluated by examining the presence of malaria parasites in the midgut of mosquitoes fed on study participants. The human-to-mosquito transmission by DSF and EH assay methods will be analyzed for potential correlation.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Currently enrolled in the PfSPZ Vaccine trial.
* Willingness to participate in the study as evidenced by signing the informed consent document, or by fingerprinting the consent document and obtaining the signature of a witness.

EXCLUSION CRITERIA:

* Refusal to participate
* Known history of abnormal reaction to mosquito bites
* Any condition that in the opinion of the investigator would jeopardize the safety or rights of a volunteer participating in the DSF or EH procedures or would render the volunteer unable to comply with the Feeding Assay Protocol.
* Pregnancy
* Any condition that in the opinion of the investigator would withdraw the volunteer from vaccine trial.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2014-07-16; Primary Completion 2014-07-16 (Actual); Study Completion 2014-07-16 (Actual)

PRIMARY OUTCOMES:
Measurement of infection/infectivity incidences | 1 year

SECONDARY OUTCOMES:
Measurement of infection intensity for a given mosquito that was fed on a given subject | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Sara A Healy, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- Malaria Research and Training Center, Bamako, Mali

REFERENCES:
- [Background] Diallo M, Toure AM, Traore SF, Niare O, Kassambara L, Konare A, Coulibaly M, Bagayogo M, Beier JC, Sakai RK, Toure YT, Doumbo OK. Evaluation and optimization of membrane feeding compared to direct feeding as an assay for infectivity. Malar J. 2008 Dec 2;7:248. doi: 10.1186/1475-2875-7-248. PMID 19055715
- [Background] Gouagna LC, Yao F, Yameogo B, Dabire RK, Ouedraogo JB. Comparison of field-based xenodiagnosis and direct membrane feeding assays for evaluating host infectiousness to malaria vector Anopheles gambiae. Acta Trop. 2014 Feb;130:131-9. doi: 10.1016/j.actatropica.2013.10.022. Epub 2013 Nov 18. PMID 24262642
- [Background] Moorthy VS, Newman RD, Duclos P, Okwo-Bele JM, Smith PG. Assessment of the RTS,S/AS01 malaria vaccine. Lancet Infect Dis. 2013 Apr;13(4):280-2. doi: 10.1016/S1473-3099(13)70047-1. Epub 2013 Mar 1. No abstract available. PMID 23454165